CLINICAL TRIAL: NCT06163521
Title: The Effect of Awareness Training Programme on School Age Children's Attitudes Towards Children With Special Needs: A Mixed Method Research
Brief Title: The Effect of Education Programme on School Age Children's Attitudes Towards Children With Special Needs
Acronym: Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, SÜMEYYE KAYA KOCAGİL, Principal Investigator, Mersin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SKaya_001
Record Dates: First submitted 2023-11-25; First posted 2023-12-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Attitude
Keywords: Special needs; Attitude; School age children
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Pre-experimental, nested design in mixed methodology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — A training consisting of 8 sessions of 40 minutes each will be applied to the children. One session will be done every week. The training will consist of activities including information, discussion and role-playing about children with special needs. The training topics consist of; Children with Special Needs Empathy Differences, Respect for Differences Contact Activity Awareness Benevolence Social Acceptance and Behaviour What can we do?

SUMMARY:
As individuals with special needs take more roles in social life and become more visible, the importance of social acceptance of individuals with special needs has increased.Especially being accepted by their peers with normal development and developing as a part of the society will reduce the burden of care in the society and enable children with special needs to lead a life worthy of human dignity.With this study, it is aimed to support children with normal development to form positive attitudes with awareness training. Qualitative and quantitative data will be used together and the attitude before and after the training will be examined descriptively.

DETAILED DESCRIPTION:
Attitudes of normally developing children towards special children may be hurtful and affect their development negatively. For this reason, by conducting an educational process in which they can develop positive attitudes, social acceptance of children with special needs can be increased, their development and psychosocial support systems can be established. Within the scope of the advocacy and health promotion role of paediatric nursing, it has the responsibility to create an environment that supports the development of children with special needs and to carry out social awareness studies. In this context, children in the school period, where attitudes, behaviour patterns and habits begin to take shape, should be supported in developing positive attitudes.In this planned study, an eight-week training process will be carried out. It is planned to reveal more comprehensive results by using qualitative and quantitative data collection methods together in the evaluation of attitude changes before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Without any disability
* Parents and siblings do not have a disability
* Have the ability to read and write in Turkish
* No child with a disability in their class
* Children aged 9-10 years attending primary school in Mersin province

Exclusion Criteria:

* With any disability
* Parents and siblings have a disability
* No ability to read and write in Turkish
* A child with a disability in their class Written, verbal consent is not obtained

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Attitudes of school children towards children with special needs ( We will use Chedoke- McMaster Attitude Scale towards Children with Disabilities.) | Before the intervention, Immediately after the intervention and one month after completion of the study.
  The scale is a Likert-type scale consisting of 31 items and is based on children's self-reports. The answers are 0 (strongly disagree), 1 (disagree), 2 (not sure), 3 (agree), 4 (strongly agree). A minimum score of 0 and a maximum score of 124 is obtained from the scale. Scores ranging from 0 to 124 points are obtained in the scale (Chedoke- McMaster Attitude Scale towards Children with Disabilities). As the score increases, children's attitudes change positively.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Yiğit, Proffessor, Study Director — Mersin University
Locations (1):
- Sümeyye Kaya Kocagil, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicek Gumus E, Oncel S. Validity and Reliability of The Chedoke-McMaster Attitudes Towards Children with Handicaps Scale in Turkey: A Methodological Study. Florence Nightingale J Nurs. 2020 Mar 6;28(1):1-12. doi: 10.5152/FNJN.2020.426719. eCollection 2020 Feb. PMID 34263180
- [Background] Alnahdi GH, Schwab S, Elahdi A, Alnahdi AH. The Positive Impact of Joint Activities on Students Attitudes Toward Peers With Disabilities. Front Psychol. 2021 Sep 8;12:690546. doi: 10.3389/fpsyg.2021.690546. eCollection 2021. PMID 34566769